CLINICAL TRIAL: NCT05417451
Title: Multi-Omics Study of the Effect and Mechanisms of Acupuncture on Psychoneurological Symptoms Among Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Hongjin Li, Assistant Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-0840
Record Dates: First submitted 2022-05-26; First posted 2022-06-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acupuncture (Experimental): All subjects will receive active acupuncture. The acupuncture intervention will consist of 10 acupuncture sessions, twice weekly for 5 weeks. There will be at least 1 day in between session.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — All participants will receive a semi-standardized acupuncture protocol (standardized points for pain, fatigue, depression, anxiety, sleep disturbance, with additional points for patient's particular pain location)

SUMMARY:
The objectives of this study to explore whether acupuncture can improve the psychoneurological symptom cluster (pain, fatigue, sleep disturbance) in survivors of breast cancer and explore biomarker changes after the acupuncture intervention. Acupuncture treatments will be provided to breast cancer survivors twice weekly for 5 weeks.

DETAILED DESCRIPTION:
The investigators will conduct the study with early stage breast cancer survivors who have completed their primary cancer treatment. They will all receive acupuncture. Treatments will be twice weekly for 5 weeks, for 30 minutes per treatment. At baseline and post-treatment, subjects will be collected blood and stool samples, complete symptom questionnaires that measure pain, fatigue, and sleep disturbance.

ELIGIBILITY:
Inclusion Criteria:

* women with histologically confirmed stage 0, I, II, or III breast cancer
* who have completed their primary cancer treatment (e.g., surgery, radiotherapy, chemotherapy) at least 3 months prior and within 5 years
* are currently receiving adjuvant endocrine therapy
* are able to read and speak English
* with self-reported pain, fatigue, sleep disturbance in the last three months and their "worst" severity rating ≥ 3 (0-10 numeric rating scale) for at least two of the three symptoms

Exclusion Criteria:

* have self-reported hospitalization for psychiatric illness within the past 2 years
* have a bleeding disorder
* physically or cognitively unable to complete the study procedures
* pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
PROMIS Pain Interference | After 10th acupuncture treatment, at 6 weeks post-baseline (study completion)
  Scores range from 4-20; higher scores indicate that pain is interfering with daily activities more
PROMIS Fatigue | After 10th acupuncture treatment, at 6 weeks post-baseline (study completion)
  Scores range from 4-20; higher scores indicate that severe fatigue
PROMIS Sleep Disturbance | After 10th acupuncture treatment, at 6 weeks post-baseline (study completion)
  Scores range from 4-20; higher scores indicate that severe sleep disturbance

SECONDARY OUTCOMES:
PROMIS Depression | After 10th acupuncture treatment, at 6 weeks post-baseline (study completion)
  Scores range from 4-20; higher scores indicate that severe depression
PROMIS Anxiety | After 10th acupuncture treatment, at 6 weeks post-baseline (study completion)
  Scores range from 4-20; higher scores indicate that severe anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago College of Nursing, Chicago, Illinois, United States